CLINICAL TRIAL: NCT02134002
Title: Dopamine Beta-hydroxylase Inhibition Induced Blunting of Dopaminergic Response to Psychostimulant Administration. A PET Exploration of the Mechanism of Action of a New Therapeutic Strategy in Cocaine Addicts
Brief Title: A PET Exploration of the Mechanism of Action of Dopamine Beta-hydroxylase Inhibition in Cocaine Addicts
Acronym: RAPID
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Too selective recrutment criteria, none eligible patients
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P121006
Record Dates: First submitted 2014-05-07; First posted 2014-05-08 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Cocaine Dependence
Keywords: cocaine; disulfiram; beta-dopamine hydroxylase
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Disulfiram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disulfiram (Experimental): disulfiram 250 mg/day
  Interventions: Drug: Disulfiram
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Disulfiram — Thirty cocaine dependant patients will be included in this study during their hospitalization for withdrawal. After the inclusion visit, they will be randomized to receive disulfiram 250 mg/day or placebo over the 15 days of their hospitalization.
  Arms: Disulfiram
Drug: Placebo — Thirty cocaine dependant patients will be included in this study during their hospitalization for withdrawal. After the inclusion visit, they will be randomized to receive disulfiram 250 mg/day or placebo over the 15 days of their hospitalization.
  Other Names: Placebo of disulfiram
  Arms: Placebo

SUMMARY:
This study represents a randomized, double blind placebo-controlled trial. Thirty cocaine dependant patients will be included in this study during their hospitalization for withdrawal. After the inclusion visit, they will be randomized to receive disulfiram 250 mg/day or placebo over the 15 days of their hospitalization. Main outcome criteria will be evaluated during two TEP imaging sessions with 11Craclopride, before and after stimulation by methylphenidate, 8 to 15 days after randomization.

DETAILED DESCRIPTION:
"Dopamine beta-hydroxylase (DHB) inhibition represents a promising approach to treating cocaine dependence. DBH is the enzyme responsible for hydroxylation of dopamine into noradrenaline. Its inhibition suppresses noradrenaline secretion. In animal studies, the efficacy of DBH inhibition in psychostimulants use could be linked to a reduced dopaminergic response, possibly in association with post synaptic dopaminergic receptor hypersensitivity. In humans, the clinical efficacy of DBH inhibition, in particular following disulfiram administration, is in the process of being established. However, its particular mode of action remains unclear: some publications suggest an increased aversive reaction to cocaine, whereas others report decreased positive effects. To date, the impact of DBH inhibition on dopaminergic response to psychostimulants has yet to be studied in humans.

This study represents a randomized, double blind placebo-controlled trial. Thirty cocaine dependant patients will be included in this study during their hospitalization for withdrawal. After the inclusion visit, they will be randomized to receive disulfiram 250 mg/day or placebo over the 15 days of their hospitalization. Main outcome criteria will be evaluated during two TEP imaging sessions with 11Craclopride, before and after stimulation by methylphenidate, 8 to 15 days after randomization. The main outcome criterion will be the variations in linkage rates of 11Craclopride in the nucleus accumbens between baseline TEP measurement and TEP measurement following administration of 20 mg of methylphenidate.

The primary objective of this trial is to show that in abstinent cocaine patients, DBH inhibition by disulfiram induces reduced dopaminergic response following methylphenidate administration. The secondary objectives of this trial are:

1. to show that methylphenidate stimulation induces less craving and more aversive responses in the disulfiram vs placebo condition;
2. to show that DBH inhibition by disulfiram elevates D2 dopaminergic receptor availability (in the absence of methylphenidate stimulation);
3. to show that the availability of D2 dopaminergic receptors (in the absence of methylphenidate stimulation) is linked to DBH activity;
4. to confirm that in abstinent cocaine patients, disulfiram reduces DBH activity vs placebo;
5. to confirm that subjects with weak DBH activity have more aversive reactions to cocaine.

Currently, disulfiram is the only drug on the market that inhibits DBH. Another more specific DBH inhibitor is currently under development. It is possible that other inhibitors could soon be developed by the pharmaceutical industry in the area of psychoactive drug addiction or other psychiatric or somatic disorders. The development of this new therapeutic approach requires a better understanding of its action mechanism.

"

ELIGIBILITY:
Inclusion Criteria:

* men aged 18 years ans less than or equal 65
* diagnosis of cocaine dependence according to DSM IV
* hospitalization for cocaine withdrawal
* ability to understand and give informed consent orally ans in writing
* affiliation to a social security
* patient with a normal ECG and normal blood pressure

Exclusion Criteria:

* Psychiatric comorbidity : psychotic disorder, manic episode , major depressive current , high suicide risk , assessed by structured interview of the Mini International Neuropsychiatric Interview
* Neurological histories: neurological deficit focused, organic cerebral disorder , epilepsy, dementia
* Severe hepatic insufficiency
* Severe renal insufficiency
* Severe respiratory
* Diabetes
* Hypersensitivity disulfiram or any of the other components
* Neuropsychological disorder
* Preexisting cardiovascular disorders
* Hypersensitivity to methylphenidate or any of the excipients
* Hyperthyroidism or thyrotoxicosis
* Glaucoma
* Pheochromocytoma
* Preexisting cerebrovascular disorders
* Patient presenting an allergy to the wheat
* HIV or HCV seropositivity
* Family or personal history of motor tics, and syndrome of Gilles Tourette
* Any disorder that may interfere with adherence to treatment
* Pharmacological treatment interfering with catecholamines
* Participation in another clinical trial or exclusion period of a previous clinical trial
* Contraindications to magnetic resonance imaging
* People under placement measure
* Hypersensitivity to any component of NIQUITIN
* Skin disorder that may interfere with the use of a transdermal patch
* Patient under treatment with irreversible inhibitors of mono- amine oxidase inhibitors (MAOIs ) , and for at least 14 days following the stop of the treatment by an IMAO.
* Diagnosis or history of bipolar disorders (affective ) episodic and severe ( type 1 )"

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Variations in linkage rates of 11Craclopride in the nucleus accumbens between baseline TEP measurement and TEP measurement following administration of 20 mg of methylphenidate. | up to 15 days after randomization
  The primary objective of this trial is to show that in abstinent cocaine patients, DBH inhibition by disulfiram induces reduced dopaminergic response following methylphenidate administration.

SECONDARY OUTCOMES:
DBH activity as measured directly, and indirectly by the DHPG / DOPAC report. | Before and after stimulation by methylphenidate, 8 to 15 days after randomization.
Measurement of craving in cocaine by a simple Likert scale. | Before and after stimulation by methylphenidate, 8 to 15 days after randomization.
Measure of aversion to cocaine by a simple Likert scale. | before and after stimulation by methylphenidate, 8 to 15 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Henri-Jean AUBIN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Paul Brousse Hospital, Villejuif, France